CLINICAL TRIAL: NCT01369888
Title: A Phase I/II Study of IL-15 Administration Following a Non-Myeloablative Lymphocyte Depleting Chemotherapy Regimen and Autologous Lymphocyte Transfer in Metastatic Melanoma
Brief Title: Use of IL-15 After Chemotherapy and Lymphocyte Transfer in Metastatic Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Closed this protocol due to autoimmune toxicity.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Steven Rosenberg, M.D., Principal investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 110170; 11-C-0170
Record Dates: First submitted 2011-06-08; First posted 2011-06-09 (Estimated); Results first posted 2015-01-27 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Metastatic Melanoma; Skin Cancer
Keywords: Immunotherapy; Cell Therapy; IL-15 Cytokine; Melanoma; Metastatic Melanoma; Skin Cancer
MeSH Terms: conditions — Melanoma; Skin Neoplasms | interventions — Cyclophosphamide; fludarabine; fludarabine phosphate; Interleukin-15

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- IL-15 following Young TIL (0.25 mcg) (Experimental): 0.25 mcg/kg/day x 10
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor Infiltrating Lymphocytes; Drug: IL-15
- IL-15 following Young TIL (0.50 mcg) (Experimental): 0.50 mcg/kg/day x 10
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor Infiltrating Lymphocytes; Drug: IL-15
- IL-15 Following Young TIL (1 mcg) (Experimental): 1 mcg/kg/day x 10
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor Infiltrating Lymphocytes; Drug: IL-15
- IL-15 Following Young TIL (2 mcg) (Experimental): 2 mcg/kg/day x 10
  Interventions: Drug: Cyclophosphamide; Drug: Fludarabine; Biological: Tumor Infiltrating Lymphocytes; Drug: IL-15

INTERVENTIONS:
Drug: Cyclophosphamide — 60 mg/m^2, intravenous (IV) (in the vein) x 2 days
  Other Names: Cytoxan
Drug: Fludarabine — 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days (days -5 to -1)
  Other Names: Fludara
Biological: Tumor Infiltrating Lymphocytes — IV over 30 minutes on day 0
  Other Names: TIL
Drug: IL-15 — IV over 30 minutes, daily for 10 days, starting 3-4 hours after the TIL infusion. (day 0 to day 9). Doses will be increased every 3-6 patients.
  Other Names: Interleukin 15

SUMMARY:
Background:

- Researchers have developed an experimental cancer treatment called cell therapy. White blood cells called lymphocytes are taken from a tumor, grown in large numbers in the lab, and then given back to the patient. Interleukin-15, given to the patient after the cells (now called Young tumor-infiltrating lymphocytes of Young TIL cells) are replaced, helps the cells to grow and boosts the immune system. This process changes your normal cells into cells that are able to recognize your tumor has been studied in the lab. These cells can destroy tumor cells in the test tube, but scientists want to see if they work inside the body.

Objectives:

-To test the effectiveness of lymphocytes drawn from tumor cells combined with interleukin-15 in treating metastatic melanoma.

Eligibility:

* Patients must be 18 - 66 years of age and have a diagnosis of metastatic melanoma.
* They will have heart and lung function tests, lab tests, and imaging procedures.
* Patients may not have conditions such as active systemic infections, blood clotting disorders, or other active major medical illnesses.
* Patients may not be pregnant or nursing.

DETAILED DESCRIPTION:
Background:

* Tumor Infiltrating Lymphocytes (TIL) can mediate the regression of bulky metastatic melanoma when administered to the autologous patient along with high-dose aldesleukin (IL-2) following a non-myeloablative lymphodepleting chemotherapy preparative regimen.
* In our analysis of factors that relate to the ability of this treatment to mediate objective responses, we have found a highly significant inverse correlation between reconstitution of cluster of differentiation 4 (CD4)+ forkhead box P3 (Foxp3) + T regulatory cells and the likelihood of achieving an objective response.
* Interleukin 2 (IL-2) administration has been shown to increase the number of T regulatory cells and in our trials we have found a direct relationship between the number of IL-2 doses and the reconstitution of patients at one week with CD4+ Foxp3 + T regulatory cells.
* Interleukin 15 (IL-15) is a strong T cell growth factor, but unlike IL-2, IL-15 is not involved in the generation and maintenance of CD4+ Foxp3 + T regulatory cells that can inhibit immune reactions.
* In pre-clinical adoptive cell transfer studies utilizing a murine melanoma model, the administration of IL-15 following adoptive cell transfer improved anti-tumor effects.

Objectives:

* The primary objective of this trial is to determine the safety, toxicity, and maximum tolerated dose of intravenous recombinant IL-15 administered as a daily intravenous bolus for 10 consecutive days in patients with metastatic melanoma who have received a lymphodepleting chemotherapy regimen and adoptive transfer of tumor infiltrating lymphocytes.
* An additional primary objective is to determine whether this combination is able to produce a modest number of clinical responses.
* The secondary objective involves the determination of the level of reconstitution of T regulatory cells in patients who receive cell transfer followed by IL-15 and to determine the pharmacokinetics of IL-15 levels in the serum following intravenous administration.

Eligibility:

* Patients greater than or equal to 18 years old with pathologically confirmed diagnosis of metastatic melanoma.
* Patients with measurable disease, absolute neutrophil count greater than 1000/mm^3 and platelet count greater than 100,000/mm^3.
* No serious comorbid conditions such as active systemic infections, coagulation disorders, or other active major medical illnesses of the cardiovascular, respiratory or immune systems.

Design:

* Patients with metastatic melanoma will undergo resection to obtain tumor for generation of autologous TIL cultures.
* Patients will receive a non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of autologous Young TIL. In the phase 1 portion of this study, patients will receive recombinant human IL-15 at doses of 0.25, 0.5, 1 or 2 micrograms per kilogram give intravenously daily for 10 days starting on the day of cell transfer. One patient will be treated at the first dose level, if this patient experiences a dose limiting toxicity (DLT), additional patients will be treated at the dose to confirm that no greater than 1/6 patients have DLT prior to proceeding to the next higher level. If 2 DLTs are encountered in this cohort, the study will be terminated. In all other cohorts, groups of three to six patients will receive recombinant human IL-15. Should a single patient experience a dose limiting toxicity due to the cell transfer at a particular dose level, additional patients will be treated at the dose to confirm that no greater than 1/6 patients have a DLT prior to proceeding to the next higher level. If a level 2 or more DLTs in 3-6 patients has been identified, three additional patients will be accrued at the next-lowest dose, for a total of 6, in order to further characterize the safety of the maximum tolerated dose prior to starting the phase 2 portion. In the phase 2 portion of this study, patients will receive a non-myeloablative lymphodepleting preparative regimen consisting of cyclophosphamide and fludarabine followed by the administration of autologous Young TIL and IL-15 at the maximum tolerated dose (MTD) established in the phase 1 portion.
* Studies will be performed to determine the reconstitution of patients with T regulatory cells and to determine the pharmacokinetics of IL-15 concentration in serum.

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Measurable metastatic melanoma with available autologous tumor infiltrating lymphocyte (TIL).
  2. Patients with 3 or less brain metastases are eligible. Note: If lesions are symptomatic or greater than or equal to 1 cm each, these lesions must have been treated and stable for 3 months for the patient to be eligible.
  3. Greater than or equal to 18 years of age and less than or equal to age 66.
  4. Able to understand and sign the Informed Consent Document
  5. Clinical performance status of Eastern Cooperative Oncology Group (ECOG) 0 or 1.
  6. Life expectancy of greater than three months.
  7. Patients of both genders must be willing to practice birth control from the time of enrollment on this study and for up to four months after receiving the preparative regimen.
  8. Serology:

     1. Seronegative for human immunodeficiency virus (HIV) antibody. (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who are HIV seropositive can have decreased immune-competence and thus be less responsive to the experimental treatment and more susceptible to its toxicities.)
     2. Seronegative for hepatitis B antigen, and seronegative for hepatitis C antibody. If hepatitis C antibody test is positive, then patient must be tested for the presence of antigen by reverse transcription polymerase chain reaction (RT-PCR) and be hepatitis C virus ribonucleic acid (HCV RNA) negative.
     3. Women of child-bearing potential must have a negative pregnancy test because of the potentially dangerous effects of the preparative chemotherapy on the fetus.
  9. Hematology:

     1. Absolute neutrophil count greater than 1000/mm^3 without the support of filgrastim.
     2. White blood cell (WBC) (> 3000/mm^3).
     3. Platelet count greater than 100,000/mm^3.
     4. Hemoglobin greater than 8.0 g/dl.
  10. Chemistry:

      1. Serum alanine aminotransferase (ALT)/aspartate aminotransferase (AST) less or equal to 2.5 times the upper limit of normal.
      2. Serum creatinine less than or equal to 1.6 mg/dl.
      3. Total bilirubin less than or equal to 1.5 mg/dl, except in patients with Gilbert's Syndrome who must have a total bilirubin less than 3.0 mg/dl.
  11. More than four weeks must have elapsed since any prior systemic therapy at the time the patient receives the preparative regimen, and patients' toxicities must have recovered to a grade 1 or less (except for toxicities such as alopecia or vitiligo).

      Note: Patients may have undergone minor surgical procedures within the past 3 weeks, as long as all toxicities have recovered to grade 1 or less or as specified in the eligibility criteria.
  12. Six weeks must have elapsed from the time of any antibody therapy that could affect an anti cancer immune response, including anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody therapy, at the time the patient receives the preparative regimen to allow antibody levels to decline.
  13. Patients who have previously received any anti-CTLA4 antibody and have documented gastrointestinal (GI) toxicity must have a normal colonoscopy with normal colonic biopsies.

EXCLUSION CRITERIA:

1. Women of child-bearing potential who are pregnant or breastfeeding because of the potentially dangerous effects of the treatment on the fetus or infant.
2. Active systemic infections, coagulation disorders or other major medical illnesses of the cardiovascular, respiratory or immune system, myocardial infarction, cardiac arrhythmias, obstructive or restrictive pulmonary disease.
3. Any form of primary immunodeficiency (such as Severe Combined Immunodeficiency Disease).
4. Concurrent opportunistic infections (The experimental treatment being evaluated in this protocol depends on an intact immune system. Patients who have decreased immune competence may be less responsive to the experimental treatment and more susceptible to its toxicities).
5. Concurrent systemic steroid therapy.
6. History of severe immediate hypersensitivity reaction to any of the agents used in this study.
7. Any patient known to have an left ventricular ejection fraction (LVEF) less than or equal to 45%.
8. In patients > 60 years old, documented LVEF of less than or equal to 45%.
9. Documented LVEF of less than or equal to 45% tested in patients with:

   1. clinically significant atrial and/or ventricular arrhythmias including but not limited to: atrial fibrillation, ventricular tachycardia, second or third degree heart block or.
   2. age greater than or equal to 60 years old.
10. Documented forced expiratory volume 1 (FEV1) less than or equal to 60% predicted tested in patients with:

    1. A prolonged history of cigarette smoking (20 pk/year of smoking within the past 2 years).
    2. Symptoms of respiratory dysfunction.

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A Rosenberg, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Thun MJ. Cancer statistics, 2007. CA Cancer J Clin. 2007 Jan-Feb;57(1):43-66. doi: 10.3322/canjclin.57.1.43. PMID 17237035
- [Background] Atkins MB, Lotze MT, Dutcher JP, Fisher RI, Weiss G, Margolin K, Abrams J, Sznol M, Parkinson D, Hawkins M, Paradise C, Kunkel L, Rosenberg SA. High-dose recombinant interleukin 2 therapy for patients with metastatic melanoma: analysis of 270 patients treated between 1985 and 1993. J Clin Oncol. 1999 Jul;17(7):2105-16. doi: 10.1200/JCO.1999.17.7.2105. PMID 10561265
- [Background] Gogas HJ, Kirkwood JM, Sondak VK. Chemotherapy for metastatic melanoma: time for a change? Cancer. 2007 Feb 1;109(3):455-64. doi: 10.1002/cncr.22427. PMID 17200963

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Protocol was closed due to autoimmune toxicity unlikely related to cells and probably related to the IL-15 injection seen in one pt and also due to the opening of additional surgery branch protocols suggesting pt accrual would not increase in this protocol. The maximum tolerated dose (MTD) was not determined and it did not enter the phase 2 stage.
Period: Overall Study
Arm/Group | IL-15 Following Young TIL (0.25 mcg) | IL-15 Following Young TIL (0.50 mcg) | IL-15 Following Young TIL (1 mcg) | IL-15 Following Young TIL (2 mcg)
Started | 1 | 2 | 0 | 0
Completed | 1 | 2 | 0 | 0
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- IL-15 Following Young TIL (10.50 mcg): 1 mcg/kg/day x 10
  Cyclophosphamide: 60 mg/m^2, intravenous (IV) (in the vein) x 2 days
  Fludarabine: 25 mg/m^2/day intravenous piggyback (IVPB) daily over 30 minutes for 5 days (days -5 to -1)
  Tumor Infiltrating Lymphocytes: IV over 30 minutes on day 0
  IL-15: IV over 30 minutes, daily for 10 days, starting 3-4 hours after the TIL infusion. (day 0 to day 9). Doses will be increased every 3-6 patients.
- Total: Total of all reporting groups
Arm/Group | IL-15 Following Young TIL (0.25 mcg) | IL-15 Following Young TIL (0.50 mcg) | IL-15 Following Young TIL (10.50 mcg) | IL-15 Following Young TIL (2 mcg) | Total
Number analyzed (Participants) | 1 | 2 | 0 | 0 | 3
Age, Categorical [Number; unit: participants]
  <=18 years | 0 | 0 |  |  | 0
  Between 18 and 65 years | 1 | 2 |  |  | 3
  >=65 years | 0 | 0 |  |  | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.0 | 38. (5.7) |  |  | 45.7 (13.9)
Gender [Number; unit: participants]
  Female | 0 | 0 |  |  | 0
  Male | 1 | 2 |  |  | 3
Ethnicity (NIH/OMB) [Number; unit: participants]
  Hispanic or Latino | 0 | 0 |  |  | 0
  Not Hispanic or Latino | 1 | 2 |  |  | 3
  Unknown or Not Reported | 0 | 0 |  |  | 0
Race (NIH/OMB) [Number; unit: participants]
  American Indian or Alaska Native | 0 | 0 |  |  | 0
  Asian | 0 | 0 |  |  | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 |  |  | 0
  Black or African American | 0 | 0 |  |  | 0
  White | 1 | 2 |  |  | 3
  More than one race | 0 | 0 |  |  | 0
  Unknown or Not Reported | 0 | 0 |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 |  |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Phase 1: Maximum Tolerated Dose (MTD) of Intravenous Recombinant IL-15 as a Daily Intravenous Bolus for 10 Consecutive Days in Patients With Metastatic Melanoma Who Have Received a Lymphodepleting Chemotherapy and ACT TIL.
Description: Intravenous recombinant IL-15 as a daily intravenous bolus for 10 consecutive days in patients with metastatic melanoma who have received a lymphodepleting chemotherapy and ACT TIL with dose escalation (i.e., dose level 1: 0.25 mcg, dose level 2: 0.50 mcg, dose level 3: 1 mcg, and dose level 4: 2 mcg) to further characterize the safety of the MTD prior to starting the phase 2 portion.
Time Frame: 2 years
Measure: Number; unit: mcg/kg/day
Arm/Group | IL-15 Following Young TIL (0.25 mcg) | IL-15 Following Young TIL (0.50 mcg)
Number analyzed (Participants) | 1 | 2
mcg/kg/day | NA — The MTD was not determined due to the autoimmune toxicity and it did not enter the phase 2 stage. | NA — The MTD was not determined due to the autoimmune toxicity and it did not enter the phase 2 stage.

2. Primary Outcome: Number of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For a detailed list of adverse events, see the adverse event module.
Time Frame: 8 months, 9 days
Measure: Number; unit: participants
Arm/Group | IL-15 Following Young TIL (0.25 mcg) | IL-15 Following Young TIL (0.50 mcg)
Number analyzed (Participants) | 1 | 2
participants | 1 | 2

ADVERSE EVENTS:
Arm/Group | IL-15 Following Young TIL (0.25 mcg) | IL-15 Following Young TIL (0.50 mcg)
Serious Adverse Events (participants affected / at risk) | 1/1 | 0/2
Other Adverse Events (participants affected / at risk) | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-15 Following Young TIL (0.25 mcg) (N=1) | IL-15 Following Young TIL (0.50 mcg) (N=2)
Autoimmune reaction (Immune system disorders) | 1 (1) | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-15 Following Young TIL (0.25 mcg) (N=1) | IL-15 Following Young TIL (0.50 mcg) (N=2)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Lymphopenia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Platelets (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1) | 0
Infection (Infections and infestations) | 1 (1) | 0
Edema: limb (Blood and lymphatic system disorders) | 1 (1) | 0
Cognitive disturbances (Nervous system disorders) | 1 (1) | 0
Psychosis (hallucinations/delusions) (Nervous system disorders) | 1 (1) | 0 — Uninvited visual images when eyes closed.
Pain (General disorders) | 1 (1) | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0
Otitis, middle ear (non-infectious) (Ear and labyrinth disorders) | 0 | 1 (1)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 0 | 1 (1)
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10e9/L) (General disorders) | 0 | 1 (1)
Rigors/chills (General disorders) | 0 | 1 (1)
Sweating (diaphoresis) (General disorders) | 0 | 1 (1)
Weight loss (General disorders) | 0 | 1 (1)
Hot flashes/flushes (Endocrine disorders) | 0 | 1 (1)
Anorexia (Gastrointestinal disorders) | 0 | 1 (1)
Constipation (Gastrointestinal disorders) | 0 | 1 (1)
Nausea (Gastrointestinal disorders) | 0 | 1 (1)
Febrile neutropenia (Infections and infestations) | 0 | 2 (2) — (fever of unknown origin without clinically or microbiologically documented infection) (ANC <1.0 x 10e9/L, fever >38.5 degrees C)
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 0 | 1 (1)
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 0 | 1 (1)
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 0 | 1 (1)
Phosphate, serum-low (hypophosphatemia) (Metabolism and nutrition disorders) | 0 | 1 (1)
Syncope (fainting) (Nervous system disorders) | 0 | 1 (1)
Pain (General disorders) | 0 | 2 (2)
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 0 | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No